CLINICAL TRIAL: NCT05622240
Title: 99mTc-MIRC213 SPECT/CT for the Detection of HER2-positive Breast Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-MIRC213
Record Dates: First submitted 2022-11-14; First posted 2022-11-18 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: SPECT/CT; HER2
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 99mTc-MIRC213 Dosimetry study (Experimental): about 6 patients were injected with 11.1-14 (MBq) per kilogram body weight of 99mTc-MIRC213 in one dose intravenously and underwent wholebody scan at 5min、20min、40min、60min、90min、120min、180min、240min, then analysis of dosimetric distribution of radiopharmaceuticals in human body by HERMES software.
  Interventions: Drug: 99mTc-MIRC213
- 99mTc-MIRC213 wholebody and SPECT/CT scan (Experimental): About 30 patients were injected with 11.1-14 (MBq) per kilogram body weight of 99mTc-MIRC213 in one dose intravenously and underwent wholebody scan 1 \2\3h later and underwent SPECT/CT scan at 2h.
  Interventions: Drug: 99mTc-MIRC213

INTERVENTIONS:
Drug: 99mTc-MIRC213 — 99mTc-MIRC213 were intravenous injected into the patients before the wholebody and SPECT/CT scans

SUMMARY:
This is an open-label single photon emission tomography/computed tomography (SPECT/CT) study to investigate the imaging performance of 99mTc-MIRC213 in breast cancer patients. A single dose of 11.1-14.8Mega-Becquerel (MBq) per kilogram body weight 99mTc-MIRC213 will be injected intravenously. Visual and semiquantitative method will be used to assess the SPECT/CT images.

DETAILED DESCRIPTION:
99mTc-MIRC213 is an nano affibody probe targeting HER2. The investigators will determine the use of 99mTc-MIRC213 SPECT/CT in the detection of HER2- positive breast cancer, and to compare its diagnostic value with routine immunohistochemistry (IHC) pathological staining. HER2 imaging, specifically to HER2 receptor expressed on malignant breast cancer cell surface, might help for targeted therapy with monoclonal antibody such as trastuzumab in breast cancer, and may improve the treatment strategy of breast cancer. The investigator will determine the use of 99mTc-MIRC213 SPECT/CT in stratifying breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients in suspicion of breast cancer by mammography or ultrasonography,and being able to provide basic information and sign the written informed consent form

Exclusion Criteria:

* The exclusion criteria included claustrophobia, pregnancy, breastfeeding, kidney or liver failure, inability to fulfill the study, and undergoing any preceding local or systemic therapies that might interfere with HER2 binding.

Max Age: 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Dosimetric distribution of radiopharmaceuticals | 2 months
  Input the data of 5-6 patients into HERMES software, and analyze the dose distribution of radioactive drugs in human body through HERMES software
Standardized uptake value | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in breast tumor will be measured. SUV were obtained by a self-made software and referring to phantom study.If the SUV value cannot be obtained, the COUNTS of target organ/background ratio between the lesion and surrounding tissues shall be used for calculation.

SECONDARY OUTCOMES:
Adverse events collection | 1 year
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, Dr, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, China